CLINICAL TRIAL: NCT02306824
Title: Berlin Cohort Study on Oral Anticoagulation in Patients With Atrial Fibrillation and Acute Ischemic Stroke
Brief Title: Berlin Atrial Fibrillation Registry
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Principal Investigator, Karl Georg Haeusler, Prof., Charite University, Berlin, Germany
Other Study IDs: EA2/052/14
Record Dates: First submitted 2014-11-30; First posted 2014-12-03 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Acute Ischemic Stroke; Atrial Fibrillation
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigator-initiated prospective multicentre hospital-based registry to uncover the proportion of self-reported anticoagulation in stroke patients with atrial fibrillation and assessing the proportion of stroke, intracranial bleeding and all-cause death in the short (at 3 months), mid-term (at 12 months) as well as long term (at 24 months) after ischemic stroke or transient ischemic attack in an unselected urban population in Germany. In addition, annual follow-up is planned yearly up to 5 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke or transient ischemic attack (with clinical deficit on admission or corresponding brain MRI lesion)
* Age ≥ 18 years
* Known atrial fibrillation or ECG recording documenting atrial fibrillation during the in-hospital stay for acute ischemic stroke or transient ischemic attack
* Written or oral informed consent
* Willingness to take part in the planned follow up examinations

Exclusion Criteria:

* Life expectancy < 1 year (before stroke)
* Assumed post-stroke life expectancy < 1 month according to stroke severity
* Chronic anticoagulation for reasons other than atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known atrial fibrillation and acute ischemic stroke or transient ischemic attack
Sampling Method: Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2014-12; Primary Completion 2017-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Patient self-reported persistence to oral anticoagulants (novel oral anticoagulants or vitamin K antagonists) in stroke patients with AF at 12 months after ischemic stroke or TIA | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl Georg Haeusler, MD, FESC, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Olma MC, Tutuncu S, Hansen K, Grittner U, Kunze C, Dietzel J, Schurig J, Dimitrijeski B, Hagemann G, Hamilton F, Honermann M, Jungehuelsing GJ, Kauert A, Koennecke HC, Mackert BM, Nabavi DG, Schmehl I, Sparenberg P, Stingele R, Voelzke E, Waldschmidt C, Zeise-Wehry D, Heuschmann PU, Endres M, Haeusler KG. Timing of oral anticoagulation in atrial fibrillation patients after acute ischaemic stroke and outcome after 3 months: results of the multicentre Berlin Atrial Fibrillation Registry. Open Heart. 2024 Sep 18;11(2):e002688. doi: 10.1136/openhrt-2024-002688. PMID 39299734
- [Derived] Tutuncu S, Olma M, Kunze C, Dietzel J, Schurig J, Fiessler C, Malsch C, Haas TE, Dimitrijeski B, Doehner W, Hagemann G, Hamilton F, Honermann M, Jungehulsing GJ, Kauert A, Koennecke HC, Mackert BM, Nabavi D, Nolte CH, Reis JM, Schmehl I, Sparenberg P, Stingele R, Volzke E, Waldschmidt C, Zeise-Wehry D, Heuschmann PU, Endress M, Haeusler KG. Off-label-dosing of non-vitamin K-dependent oral antagonists in AF patients before and after stroke: results of the prospective multicenter Berlin Atrial Fibrillation Registry. J Neurol. 2022 Jan;269(1):470-480. doi: 10.1007/s00415-021-10866-2. Epub 2021 Oct 31. PMID 34718884